CLINICAL TRIAL: NCT00473044
Title: An Intervention to Increase Physical Activity Among African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Obidiugwu Kenrik Duru, MD, MS, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0085; R01AG024460 (NIH)
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Sedentary Lifestyle; Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Sisters in Motion

SUMMARY:
The purpose of this study is to investigate whether a faith-based curriculum delivered in small groups, and emphasizing goal setting along with mutual responsibility, increases physical activity.

DETAILED DESCRIPTION:
Sedentary lifestyles are common among older adults in the United States, especially among minority women. Regular physical activity in older adults has been shown to prevent falls, maintain functional status, prevent both dementia and osteoporosis, and decrease mortality. A review of the literature has shown that current research approaches using exercise classes as the only means of behavior change are ineffective and do not produce long-term sustainable improvement. This study is testing a culturally appropriate behavior modification intervention using 1) group prayer, 2) the development of social support and mutual responsibility for exercise, and 3) group problem solving activities to increase aerobic and strength-related activities among older African American women.

Participants randomized into the intervention arm receive a 45-minute curriculum session and a 45 minute exercise class, while those randomized into the control arm receive a 45 minute session of interactive lectures on unrelated health topics along with the 45 minute exercise class. The exercise class includes both aerobic exercise and strength training using hand-held weights.

Data is collected from pedometers worn by participants, as well as from questionnaires before and after the intervention. Blood pressure, weight, and cholesterol are measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 60 years
* Female
* African American

Exclusion Criteria:

* Use of walker for ambulation
* Positive response on a modified Physical Activity Readiness Questionnaire, indicating potential risk of engaging in activity
* Withdrawal by primary physician

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in weekly steps walked as measured by pedometer | 10 weeks and 6 months

SECONDARY OUTCOMES:
Change in weekly metabolic equivalents expended in physical activity | 10 weeks and 6 months
Change in blood pressure, weight, and low-density lipoprotein (LDL) cholesterol | 10 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Obidiugwu Kenrik Duru, MD, Principal Investigator — David Geffen School of Medicine, University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Dunn AL, Blair SN. Translating evidenced-based physical activity interventions into practice. The 2010 challenge. Am J Prev Med. 2002 May;22(4 Suppl):8-9. doi: 10.1016/s0749-3797(02)00432-4. No abstract available. PMID 11985931
- [Background] American College of Sports Medicine. Physical activity programs and behavior counseling in older adult populations. Med Sci Sports Exerc. 2004 Nov;36(11):1997-2003. doi: 10.1249/01.mss.0000145451.08166.97. PMID 15514518
- [Background] Brawley LR, Rejeski WJ, King AC. Promoting physical activity for older adults: the challenges for changing behavior. Am J Prev Med. 2003 Oct;25(3 Suppl 2):172-83. doi: 10.1016/s0749-3797(03)00182-x. PMID 14552942